CLINICAL TRIAL: NCT00073788
Title: Wounded Spirits, Ailing Hearts: Post-Traumatic Stress Disorder and Cardiovascular Disease in Indians
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 03-1028; R01HL073824 (NIH)
Record Dates: First submitted 2003-12-08; First posted 2003-12-10 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with PTSD: Subjects will be American Indian, between the ages of 18-68. Approximately 66% will be female, 33% male, which conforms to the distribution of PTSD in this population. Study group subjects will be PTSD positive. Overt CVD is exclusionary.
  Interventions: Procedure: PET Scans
- Control Group: Subjects will be American Indian, between the ages of 18-68. Approximately 66% will be female, 33% male, which conforms to the distribution of PTSD in this population. Control subjects will be PTSD negative. For both groups: overt CVD is exclusionary.
  Interventions: Procedure: PET Scans

INTERVENTIONS:
Procedure: PET Scans — PET Scan to look for coronary flow reserve, heart rate variability, and carotid ultrasound measures (mean intermediate thickness of the far fall of the carotid artery).

SUMMARY:
To evaluate Post-Traumatic Stress Disorder as a risk factor for cardiovascular disease in American Indians.

DETAILED DESCRIPTION:
BACKGROUND:

Post-Traumatic Stress Disorder (PTSD) is a unique psychiatric condition characterized by a persistent maladaptive reaction resulting from exposure to a stressful traumatic event(s). In the United States general population PTSD has a lifetime prevalence of 5 percent in men and 10 percent in women. PTSD is known to produce alternations in the central and autonomic nervous system and hormonal dysregulation. However, little is known about the long-term consequences of PTSD on the cardiovascular system. PTSD is a common disorder among reservation dwelling American Indians with a life-time prevalence of 12 percent in men and 23 percent in women. Similarly, cardiovascular disease (CVD), has emerged as a major health problem in American Indians during the past decade.

DESIGN NARRATIVE:

The study examines the relationship between PTSD and cardiac function in a population-based sample of American Indians. The technical aims of this study involve: 1) the identification of American Indian men and women ages 18-52 who have a lifetime history of PTSD and are free from overt CVD; 2) the selection of an age-, sex-, and tribe-matched comparison group of American Indians who have no history of PTSD and are free from known CVD; 3) a comprehensive lifestyle and clinical evaluation of the PTSD and non-PTSD groups to assess CVD risk factors such as smoking, exercise, obesity, blood pressure, concentrations of blood lipids, and inflammatory and thrombogenic factors; and 4) a set of non-invasive tests of subclinical CVD and other measures of CVD risk. These tests include positron emission tomography (PET) myocardial perfusion imaging to examine coronary flow reserve, high-resolution ultrasound of the carotid arteries to measure carotid intima-media thickness, high-resolution ultrasound of the brachial artery to determine flow-mediated vasodilation, and ambulatory electrocardiographic monitoring, to assess heart rate variability (HRV). With these data, the study addresses the specific aims, which are: 1) to determine whether individuals with PTSD, compared with those without PTSD, show greater evidence of subclinical CVD, including a lower coronary flow reserve, increased carotid intimamedia thickness, and reduced forearm flow-mediated vasodilation; 2) to ascertain whether HRV is lower in individuals with PTSD compared to those without PTSD; and 3) to investigate the role of lifestyle (e.g., smoking, alcohol use, exercise, obesity), cultural (e.g., acculturation, religiosity), and biological (e.g., blood pressure, blood lipid and glucose concentrations) mediators in the relationship of PTSD with coronary flow reserve and HRV.

ELIGIBILITY:
Inclusion criteria

* be 18 years of age or older;
* not be pregnant, or breastfeeding;
* be free of heart disease when they participated in the American Indian Services Utilization, Psychiatric Epidemiology, Risk and Protective Factors Project (AI-SUPERPFP); or change in PTSD status from time of participation to completion of 2nd stage screening;
* have no medical issues that interfere with the PET imaging such as unstable angina, myocardial infarction in the past week, severe obstructive lung disease, decompensated heart failure; severe coronary disease, severe stroke, or other medical conditions that would make it unsafe for them to travel and complete the protocol (e.g., not be on dialysis);
* not be taking any medications such as theophylline or aminophylline or oral steroids (e.g. prednisone);
* participants who use inhalers or nebulizers will be asked to use the inhalers or nebulizers in Denver on their regular schedule. If they are able to administer these treatments themselves on their regular schedule, they are eligible to be brought to Denver, assuming other eligibility criteria are met.
* and not have any conditions or devices, like claustrophobia that would interfere with the heart imaging process.
* not be using alcohol or any illegal substances during Denver visit and examination period.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: American Indian people with, and without, PTSD
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2003-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
coronary flow reserve | study visit
  Measured by PET Scan. For coronary flow reserve, we will mainly focus on the overall measure of coronary flow reserve (as opposed to regional analysis), since this is thought to be appropriate for detection of early coronary disease.
Heart Rate Variation (HRV) | study visit
  Measured by PET Scan. The main outcome for HRV will be the high frequency power.
carotid intima-media thickness | study visit (PET scan)
  Measured by PET Scan and ultrasound. The main outcome of the carotid ultrasound will be the mean intima-media thickness on the far wall of the common carotid artery.

CONTACTS AND LOCATIONS:
Overall Officials: Spero M. Manson, PhD, Principal Investigator — University of Colorado, Denver